CLINICAL TRIAL: NCT05564208
Title: A Phase I, Open-Label, Randomised, Balanced, Single-Dose, Two-Period, Two-Sequence Crossover-Design Study to Evaluate Effects of Food on the Bioavailability of 80 mg Elafibranor (IPN60190) To-be-marketed Tablet Formulation After Single Oral Administration in Healthy Adult Participants
Brief Title: A Study to Evaluate the Effect of Food on the Level of Circulating Elafibranor in Healthy Participants After Intake of a Single Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CLIN-60190-452; 2022-001883-91 (EudraCT Number)
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Healthy Participants
Keywords: Pharmacokinetics; Elafibranor
MeSH Terms: interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elafibranor Fasting then Elafibranor fed (Experimental): Participants will receive Elafibranor 80 mg in Fasting State on Day 1 of Period 1 followed by a washout period of a maximum of 28 days. Participants will then receive Elafibranor 80 mg in Fed State on Day 1 of Period 2.
  Interventions: Drug: elafibranor
- Elafibranor Fed then Elafibranor fasting (Experimental): Participants will receive Elafibranor 80 mg in Fed State on Day 1 of Period 1 followed by a washout period of a maximum of 28 days. Participants will then receive Elafibranor 80 mg in Fasting State on Day 1 of Period 2.
  Interventions: Drug: elafibranor

INTERVENTIONS:
Drug: elafibranor — Oral Tablet
  Other Names: GFT505; IPN60190
  Arms: Elafibranor Fasting then Elafibranor fed
Drug: elafibranor — Oral Tablet
  Other Names: GFT505; IPN60190
  Arms: Elafibranor Fed then Elafibranor fasting

SUMMARY:
This study will evaluate the effects of food on how much test drug is able to access the circulation and reach the target area (known as bioavailability).

The test drug, elafibranor (IPN60190), is in development for the treatment of primary biliary cholangitis (PBC).

PBC is a rare, long-term autoimmune disease of the liver. An autoimmune disease occurs when the immune (defence) system treats healthy parts of the body as if they were foreign and attacks them.

This study will be in healthy volunteers, so this trial is not to test if the drug helps to improve health.

ELIGIBILITY:
Inclusion Criteria :

* Willingness to remain at the clinic for the required duration and willingness to return to the clinic for the follow-up evaluation as specified in the protocol
* Healthy participants as determined by medical evaluation at the screening visit including medical history, physical examination, laboratory tests, electrocardiogram (ECG) and vital signs monitoring
* Laboratory parameters within the normal range of the laboratory (haematological, blood biochemistry, urinalysis) at screening and baseline visit of each period. Individual values out of the normal range can be accepted if judged not clinically significant by the investigator
* Normal electrocardiogram (ECG) recording on a 12-lead ECG at screening and baseline visit of each period:

  * 120≤PR≤220 ms,
  * QRS<110 ms,
  * QTcF≤430 ms for male and
  * ≤450 ms for female,
* No evidence of sinus node automaticity or abnormal conduction, or rhythm disorders of concern, except as considered not clinically significant by the investigator. Out-of-range values that are not clinically significant (as determined by the investigator) may be repeated twice during screening and baseline visits of each period and the participant may be enrolled if at least one repeated value is within the range noted above.
* Normal blood pressure (BP) and heart rate (HR) at screening and baseline visits of each period after 5 minutes in supine position:

  * 90 mmHg≤systolic blood pressure (SBP)≤145 mmHg,
  * 50 mmHg≤diastolic blood pressure (DBP)≤90 mmHg,
  * 45 bpm≤HR≤90 bpm,
* For these parameters, out-of-range values that are not clinically significant (as determined by the investigator) may be repeated twice during screening and baseline visits of each period and the participant may be enrolled if at least one repeated value is within the range noted above.
* Body weight not below 55 kg and body mass index (BMI) within the range 20.0 kg/m^2 and 28.0 kg/m^2 (inclusive) at screening.
* Contraception/barrier requirements: Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding at screening, is willing not to become pregnant during the study, and is willing to follow applicable protocol requirements related to this. Male participants are eligible to participate if they agree to follow applicable protocol requirements related to contraception.

Exclusion Criteria :

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, haematological or neurological disorders capable of significantly altering the absorption, metabolism or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Lymphoma, leukaemia or any malignancy within the past 5 years except basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years prior to screening
* Breast cancer within the past 10 years at screening
* Major surgery within 28 days prior to screening
* Past or intended use of over the counter (OTC) or prescription medication (including herbal medications or vitamin supplements, nutritional supplements, herb-containing drug preparations (including Chinese medicines)) within 14 days or 5 half-lives of the drug (whichever is longer) prior to dosing. Exceptions are oral contraception/hormone replacement therapy for females and paracetamol/acetaminophen at doses of ≤2 g/day.
* Any vaccination during the 4 weeks before randomisation or planned during the clinical study
* Use of any medications within 3 months that may interfere with absorption, distribution, metabolism or excretion of the study intervention, or any medication that may result in induction or inhibition of microsomal enzymes.
* Plasma donation within 14 days of the screening or any blood donation/ blood loss >450 mL during the last 30 days before screening. Blood and/or plasma should not be donated until 30 days after last study intervention.
* Current enrolment or past participation within the last 3 months (or 5 half-lives, whichever is longer) before signing of consent in any other clinical study involving an investigational study intervention or any other type of medical research.
* Participant who would receive more than 4500 Euro as indemnities for participation in biomedical research within the last 12 months, including the indemnities for the present study.
* Presence of hepatitis B surface antigen (HBsAg) at screening
* Positive hepatitis C antibody test result at screening. NOTE: Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled if a confirmatory negative hepatitis C ribonucleic acid (RNA) test is obtained and sustained viral response can be documented
* Positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention. NOTE: Test is optional and participants with negative hepatitis C antibody test are not required to also undergo hepatitis C RNA testing
* Positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) antigen test result at screening or during the study
* Positive drugs of abuse/alcohol screen at screening and baseline visit of each period
* Positive human immunodeficiency virus (HIV) antibody test at screening
* Consumption of other foods or beverages (e.g. red wine, Seville oranges, grapefruit orgrapefruit juice (including pomelos, exotic citrus fruits, grapefruit hybrids, or fruit juices)) that may affect drug-metabolising enzymes or transporters from 7 days prior to dosing until the end of each study period
* Inability to abstain from caffeine- or xanthine-containing products (e.g. coffee, tea, cola drinks and chocolate) for 24 hours before dosing until after collection of the final PK sample in each period
* Any history or suspicion of alcohol abuse (alcohol consumption >40 g/day). Inability to abstain from alcohol for 24 hours before each period and until after the last sample from each period is collected
* History of illicit drug abuse within the last 12 months
* Sensitivity to any components of the study intervention or other allergy that, in the opinion of the investigator, contraindicates participation in the study, including lactose intolerance
* Inability to abstain from intensive muscular effort. Participants should not engage in any strenuous activity from 72 hours prior to admission to the clinical unit until after their EOS visit
* Smoker. Smoking or use of tobacco or nicotine-containing products within 3 months prior to or during the study. Status will be confirmed with a urine cotinine at screening and at baseline visits of each period
* Had been on a diet incompatible with the on-study diet (i.e. unusual meal habits, special diet requirements or unwillingness to eat the food provided in the study, e.g. vegetarian nor vegan), in the opinion of the investigator or designee, within the 30 days prior to the first dosing and throughout the study
* Venous status at forearm or dorsal hand making it difficult to insert a venous peripheral catheter
* Vulnerable subjects, e.g. kept in detention, protected adults under guardianship, trusteeship or committed to an institution by governmental or juridical order

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-14 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of Elafibranor: Area Under the Plasma Concentration Time Curve From Zero to the Last Quantifiable Concentration (AUC0-t) | Day 1 up to Day 10
  AUC0-t will be recorded from the PK blood samples collected.
PK of Elafibranor: Area Under Plasma Concentration Time Curve From Zero to Infinity (AUC0-∞) | Day 1 up to Day 10
  AUC0-∞ will be recorded from the PK blood samples collected.
PK of Elafibranor: Maximum Observed Plasma (peak) Drug Concentration (Cmax) | Day 1 up to Day 10
  Cmax will be recorded from the PK blood samples collected.

SECONDARY OUTCOMES:
PK of Elafibranor's Metabolite GFT1007: Area under the Plasma Concentration Time Curve From Zero to the Last Quantifiable Concentration (AUC0-t) | Day 1 up to Day 10
  AUC0-t will be recorded from the PK blood samples collected.
PK of Elafibranor's Metabolite GFT1007: Area Under Plasma Concentration Time Curve From Zero to Infinity (AUC0-∞) | Day 1 up to Day 10
  AUC0-∞ will be recorded from the PK blood samples collected.
PK of Elafibranor's Metabolite GFT1007: Maximum Observed Plasma (peak) Drug Concentration (Cmax) | Day 1 up to Day 10
PK of Elafibranor and its Metabolite GFT1007: Terminal Elimination Half-life (t1/2) | Day 1 up to Day 10
  t1/2 will be recorded from the PK blood samples collected.
PK of Elafibranor and its Metabolite GFT1007: Time to Maximum Observed Drug Concentration (Tmax) | Day 1 up to Day 10
  Tmax will be recorded from the PK blood samples collected.
PK of Elafibranor and its Metabolite GFT1007: Terminal Elimination Rate Constant (λz) | Day 1 up to Day 10
  tlag will be recorded from the PK blood samples collected.
PK of Elafibranor and its Metabolite GFT1007: Terminal Elimination Rate Constant (λz) | Day 1 up to Day 10
  λz will be recorded from the PK blood samples collected.
PK of Elafibranor and its Metabolite GFT1007: Total Body Clearance (Cl/F) | Day 1 up to Day 10
  Cl/F will be recorded from the PK blood samples collected.
PK of Elafibranor and its Metabolite GFT1007: Volume of distribution (Vd/F) | Day 1 up to Day 10
  Vd/F will be recorded from the PK blood samples collected
Percentage of Participants With Treatment Emergent Adverse Event (TEAEs) and Adverse Events of Special Interest (AESIs) | Baseline up to Day 21
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AESIs are AEs that may not be serious but are of special importance to a particular drug or class of drugs
Percentage of Participants With Clinically Significant changes in Laboratory Parameters (blood chemistry, hematology and coagulation) | Baseline up to Day 21
  Percentage of participants with clinically significant change in laboratory parameters (blood chemistry, hematology and coagulation) will be reported. The clinical significance will be decided by the investigator
Percentage of Participants With Clinically Significant Changes in Vital Signs | Baseline up to Day 21
  Percentage of participants with clinically significant changes in Vital Signs will be reported. The clinical significance will be decided by the investigator.
Percentage of Participants with Clinically Significant Changes in 12-lead Electrocardiogram (ECG) Readings | Baseline up to Day 21
  Percentage of participants with clinically significant changes in ECG readings will be reported. The clinical significance will be decided by the investigator.
Percentage of Participants With Clinically Significant Changes in Physical Examination | Baseline up to Day 21
  Percentage of participants with clinically significant changes in physical examination findings will be reported. The clinical significance will be decided by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Ipse Medical Director, Study Director — Ipsen
Locations (1):
- BIOTRIAL, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2024/02/14114115/Study-CLIN-60190-452-Elafibranor-food-effect-study.pdf